CLINICAL TRIAL: NCT00149344
Title: Vertical Scar Versus Inferior Pedicle Reduction Mammoplasty: A Randomized Controlled Trial and Cost-Utility Analysis
Brief Title: Vertical Scar Versus Inferior Pedicle Reduction Mammoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Society of Plastic Surgeons (Other)
Responsible Party: Dr. Achilleas Thoma, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-2447
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Breast Hypertrophy
Keywords: cost-utility analysis;; breast reduction;; vertical scar mammoplasty;; pedicle reduction mammoplasty
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Vertical scar versus inferior pedicle reduction mammoplasty — Vertical Scar Reduction Mammoplasty Inferior Pedicle Reduction Mammoplasty

SUMMARY:
Main research question: Is vertical scar reduction mammoplasty superior when compared to inferior pedicle reduction mammoplasty in terms of patient quality of life and cost-effectiveness?

Why is this research important?: There is on-going controversy among plastic surgeons as to the superiority of one technique (vertical scar mammoplasty versus inferior pedicle reduction mammoplasty) over the other in terms of patient health related quality of life and health care resource utilization.

What is being studied?: We are studying (comparing) two surgical procedures for breast reduction mammoplasty (vertical scar mammoplasty versus inferior pedicle reduction mammoplasty).

DETAILED DESCRIPTION:
Breast reduction is one of the most common procedures performed by plastic surgeons. Because it is common and in most jurisdictions requires at least one day of hospital stay, it consumes considerable health care resources. Although multiple techniques have been reported, the two top competing techniques used in North America are the inferior pedicle technique and the vertical scar technique. There is on-going controversy as to the superiority of one technique over the other in terms of patient satisfaction and health care resource utilization. In the last few years, third party payers have been concerned with the unnecessary consumption of scarce health care resources due to the variation of practice mostly influenced by surgeon preferences rather than valid evidence.

The purpose of this study is to test the hypothesis that Vertical Scar Reduction Mammoplasty (VSR) is superior to the Inferior Pedicle Reduction Mammoplasty (IPR) in terms of patient health-related quality of life (HRQL). Health related quality of life will be measured by the Health Utilities Index Mark 2/3 (HUI) providing the outcome, quality adjusted life years (QALYs) and the Breast Reduction Assessment Value and Outcomes (BRAVO) instruments. The BRAVO instruments consist of a set of separate instruments including the Short Form 36 (SF-36), the Multidimensional Body Self Relations Questionnaire Appearance Assessment (MBSRQ-AS), and the Breast Related Symptoms Questionnaire (BRSQ). The MBSRQ-AS provides a measure of self-evaluation of appearance, and the BRSQ measures the breast symptom score. Secondly, we will test whether the VSR is a more cost-effective procedure. If the hypothesis is confirmed that the VSR technique is more cost-effective, then there will be compelling evidence to adopt it. Regardless of whether VSR is found to be cost-effective, the plastic surgery community, third party payers, and patients will be informed about the results.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from breast hypertrophy
* Patients who received OHIP approval for reduction mammoplasty
* Candidate for both surgical procedures
* Patient is willing to complete quality of life questionnaires and follow up
* Patient will provide informed consent

Exclusion Criteria:

* Unilateral Breast Hypertrophy
* Patients under the age of 18 years
* Inability to complete questionnaires due to language problems
* Bilateral mastopexy (breast lift)
* Previous breast reduction surgery
* Patients who will require greater than 1000 grams to be removed from either breast (to be assessed by the Archimedes principle* preoperatively; patients who by the Archimedes principle displace 1400 cc of volume will be excluded from the study)
* Pre-operative radiation after lumpectomy
* If another procedure is to be "piggy backed' to the reduction mammoplasty (e.g. liposuction to breast or elsewhere, abdominoplasty, etc)

  * The Archimedes principle is as follows: In the privacy of her bathroom the patient will immerse each breast separately into a large pot filled to the brim with tap water. The breast will displace some of the water which will be collected into another larger container e.g. plastic dish pan placed underneath the pot. The patient will be asked to measure the volume of the displaced water in ml. The volume that will be displaced will approximate the weight of the breast. The measurement will be done 3 times and the average for each breast will be recorded.

(The surgeon will explain this principle only to those patients where there is uncertainty whether the resection will exceed 1000 grams. For the rest of the patients this is not necessary.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2005-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (utilities and disease specific) | 1 Year

SECONDARY OUTCOMES:
Health care resource utilization as well as out-of-pocket expenses by patients and caregivers. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Achilleas Thoma, MD MSc FRCSC, Principal Investigator — McMaster University / St. Joseph's Healthcare
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Thoma A, Kaur MN, Tsoi B, Ziolkowski N, Duku E, Goldsmith CH. Cost-effectiveness analysis parallel to a randomized controlled trial comparing vertical scar reduction and inverted T-shaped reduction mammaplasty. Plast Reconstr Surg. 2014 Dec;134(6):1093-1107. doi: 10.1097/PRS.0000000000000751. PMID 25255113